CLINICAL TRIAL: NCT00855881
Title: A Trial of Metronomic Chemotherapy With Tegafur/Uracil for Patients With Locally Advanced (Stage III~IVB) Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Metronomic Chemotherapy With Tegafur/Uracil for Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Group of Head and Neck Cancer, Mackay Memorial Hospital, Taipei, Mackay Memorial Hospital, Taipei
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 376
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2010-08

CONDITIONS: Head and Neck Cancer
Keywords: adjuvant chemotherapy for head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): Treated with tegafur-uracil for 1 year
  Interventions: Drug: tegafur-uracil

INTERVENTIONS:
Drug: tegafur-uracil — tegafur-uracil 1 cap, bid for 1 year
  Other Names: UFUR

SUMMARY:
It is the investigators understanding that the combination of clinical trial with laboratory cellular/molecular assay is relevant to the current promising mainstream, the translational research. The design of this trial fulfills this concept and would be a good example conducting in Mackay Memorial hospital.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) (excluding nasopharyngeal cancer) accounts for 4% to 5% of the cancer incidence in Taiwan.1 Localized disease is curable by surgery and irradiation. Two-thirds of patients present with advanced stages of the disease (stage III and IV), and are treated with multimodality therapy, including surgery, radiation and chemotherapy. Despite the achievement of complete responses in patients who receive multimodality therapy, however, recurrences might occur in some of patients within two years after multimodality therapy.

HNSCC has been regarded as a chemosensitive tumor since the early 1980s.Cisplatin-based combination therapy with fluorouracil (5-FU) is the most common chemotherapy regimen for patients with HNSCC. Concomitant chemoradiotherapy (CCRT) is conceptually supported by the natural history of head and neck cancer, which indicates a primary need to improve locoregional therapy and only a secondary need to improve systemic therapy. CCRT has frequently been studied in inoperable patients or in those with unresectable disease4. Several recent studies and meta-analyses have indicated superior locoregional control and/or survival rates after CCRT when compared with radiotherapy alone3-12.

"Two similar, large-scale, prospective randomized independent trials designed by the European Organization for Research and Treatment of Cancer (EORTC) and the Radiation Therapy Oncology Group (RTOG) were conducted to evaluate the role of concurrent administration of cisplatin with radiation in the postoperative treatment of high-risk head and neck tumors. The EORTC (#22931) 29 study revealed that combination therapy was more efficacious than radiotherapy alone in patients with locally advanced head and neck cancer and that the treatment did not cause an undue number of late complications. The RTOG (#9501)30 trial found that postoperative CCRT significantly improved the rates of local and regional control and disease-free survival in high-risk patients with resected head and neck cancer; however, the combined treatment was associated with a substantial increase in adverse effects.

Multimodality therapy may achieve higher complete response rate for patients with locally advanced HNSCC, however, patients still face high recurrent rate that might decrease survival time. For these reasons, the development of reliable methods (for example) and metronomic therapy to prevent relapse at locally advanced setting may improve the outcome of treatment.

Uracil-tegafur (UFT), an oral fluoropyrimidine prodrug, is available commercially in Japan and in several other countries. It is composed of 1-(2-tetrahydrofuryl)-5-fluorouracil (5-FU) (FT; also ftorafur or tegafur) and uracil in a molar ratio of 1:4. FT is readily absorbed through the gut without degradation and is converted in the liver to 5-FU and subsequently degraded to 2-fluoro-b-alanine. Thus, UFT shares the chemotherapeutic mechanism of action of 5-FU. The 5-FU metabolite FdUMP binds and inhibits the enzymatic activity of thymidylate synthase (TS), thereby inhibiting DNA synthesis.13-17 Uracil strongly inhibits the degradation of 5-FU to 2-fluoro-b-alanine by competitive inhibition of dihydropyrimidine dehydrogenase (DPD), the rate-limiting enzyme in the metabolism of 5-FU.18,19 This alteration of 5-FU disposition seems to be tumor selective. When taken orally, UFT and FT give a comparable distribution of 5-FU in blood and other normal tissues, but UFT results in 5-10 times greater distribution of 5-FU in tumors.20 Co-administration of uracil and/or FT, therefore, enhances the anti-tumor activity of FT.21 The cytotoxic effects of 5-FU (and, thus, FT) can be enhanced markedly if sufficient amounts of reduced folate cofactor, such as leucovorin (LV), are present. Cellular folate pools are considered an important biochemical determinant of FdUMP enzyme binding.22-28 One basic study has shown that in mice bearing RENCA tumors, tegafur/uracil treatment resulted in significant prolongation of their life span, which was associated with the inhibition of angiogenesis. This should be recomposed. For example, "Tegafur/uracil treatment of mice with RENCA tumors has been shown to inhibit angiogenesis, leading to a significant prolongation of life span.Two metabolites of tegafur/uracil, namely, GHB33,34 and GBL were found to be responsible for these effects. In another study, the formation of cancer vasculature, essential for the initiation of metastasis and the inhibition of tumor angiogenesis, is one of the targets in tumor dormancy therapy. The efficacy of tegafur/uracil in postoperative adjuvant chemotherapy has been demonstrated in several clinical trials. The basic data from these studies indicate a possible contribution of the anti-angiogenic activity of tegafur/uracil to its overall anti-tumor activity, which until now has been thought to be mediated by the cytotoxic effects of 5-FU. Thus, tegafur/uracil seems to be particularly useful in a chronic postoperative adjuvant chemotherapy regimen to control metastasis.

Lam et31al. conducted a prospective randomized study of post-operative chemotherapy with levamisole and UFT for treatment of head and neck carcinoma. A trend towards better distant control in post-operative oral chemotherapy was observed. The side effects were minimal. Masato Fujii also reported that adjuvant chemotherapy with UFT was efficacious for treating maxillary sinus carcinoma. The 5-year survival was 76.2% for the UFT group and 17.9% for the control group32.

Metronomic chemotherapy refers to the close, regular administration of a chemotherapeutic drug, over prolonged periods, with no extended drug-free break periods38. As such, it is a form of "dose dense" chemotherapy but differs from most forms of the latter in several ways35,36. First, it is not "dose intense" when the goal remains to deliver high, toxic levels of drug over shorter periods of time. Second, because metronomic regimens are much less toxic, they do not usually require supportive growth factor, or other supportive care measures39,40. Metronomic chemotherapy can thus be viewed as a form of efficiently, low dose, and long term 'maintenance' chemotherapy that can be used on its own36,38, or more importantly, combined with long-term biologic targeted therapies, especially with antiangiogenic drugs such as anti-VEGFR-2 antibodies41 or small molecule multi-targeted VEGFR-2 antagonist receptor tyrosine kinase inhibitors42. It can also be integrated with standard MTD-type (maximum tolerated dose) chemotherapy where brief courses of such therapy, 'upfront', is followed by long-term maintenance metronomic chemotherapy combined with concurrent targeted therapies41,42, called "chemo-switching"40. The advantages of metronomic chemotherapy include reduced acute toxicities, such as high grade myelosuppression, vomiting, nausea, and mucotitis, 39,40 and sometimes surprisingly good activity against drug resistant tumors38, reduced costs when using off patent chemotherapeutic drugs, and increased convenience when using oral drugs that can be taken at home36,39. These potential advantages could be useful for long term adjuvant therapy of early stage cancers, e.g. long-term daily oral administration of a drug such as UFUR(UFT; a 5-FU prodrug) for 1~2 years with no breaks43,45,46,50.

The reason why standard chemotherapy, using a maximum tolerated dose (MTD), separated by long 2-3 week drug-free break periods is not as effective as an antiangiogenic treatment regimen is that the damage inflicted upon the dividing endothelium cells of the tumor is largely reversed during the extended drug-free break periods, perhaps by a massive hemopoiesis-like mobilization ('rebound') of CEPs which then home to damaged tumor endothelium and set about repairing the damage44. Thus shortening the break periods is critical to ensure that the repair process is prevented or minimized38. This in turn requires relatively low doses of drug to be used38.

The anti-tumor effects of single versus two chemotherapeutic drug combinations, dosed and administered in a metronomic fashion, i.e., daily (by oral delivery) in a model of advanced high volume (end stage) visceral metastatic disease where therapy is initiated in terminal stages of disease47.

Metronomic chemotherapy regimens combined with an antiangiogenic drug have moved into phase II clinical trial testing both in the adjuvant and metastatic settings. Some interim results of phase II clinical trials involving metastatic breast cancer or advanced, recurrent ovarian cancer looked extremely promising48,49,50. Ongoing, planned or recently completed phase II clinical trials of metronomic chemotherapy combined with an agent such as bevacizumab or thalidomide should indicate whether or not this treatment strategy is promising in the treatment of metastatic and/or early stage human cancer.

Although when low-dose cytotoxic drugs combined with targeted agents may have potential benefits as explained previously. There remain several significant challenges that must be overcome to increase the success in the clinical setting. Foremost among these is the current empiricism associated with trying to determine the optimal dose and schedule for administration of chemotherapeutics. The challenge lies in finding the smallest dose that will control the growth of target cells and then the most frequent dosing that will maximize this control. the discovery and application of functional surrogate markers might be one of the solutions to overcome the problem of metronomic-dose determination, such as determining the So, detecting changes in levels of circulating TSP1 levels in serum or plasma after administration of various low doses of chemotherapeutics might be useful in determining the optimal low dose for a drug such as cyclophosphamide51.

In addition to TSP1 level, the most important approach in determining the optimal metronomic low dose for a given metronomic chemotherapy regimen is evaluation of the activities of CEPs or circulating endothelial cells (CECs). As previously discussed, CEPs mobilization from the bone marrow into the peripheral circulation is strongly inhibited by low-dose cyclophosphamide, as is CEP viability52. It might be conferred that there could be a direct relationship between the relative efficacy of different (low) doses of metronomic chemotherapy and the ability of these doses to reduce levels of CEPs in the peripheral circulation. In a study by Shaked et al., using 4 distinct metronomic chemotherapy regimens in 4 different preclinical tumor models to establish optimal biological dose (OBD) without causing excessive toxicity demonstrated that the OBDs in each tumor models were strikingly correlated with the maximum reduction in CEPs53. The results of this study suggested that these results suggested that CEPs may serve as a pharmacodynamic biomarker to determine the OBD of metronomic chemotherapy regimens.

It is our understanding that the combination of clinical trial with laboratory cellular/molecular assay is relevant to the current promising mainstream, the translational research. The design of this trial fulfills this concept and would be a good example conducting in Mackay Memorial hospital.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-nasopharyngeal head and neck squamous cell carcinoma
* Complete response(CR) to previous treatment
* White blood cell (WBC) count greater than 3,000/mm3 and absolute neutrophil count (ANC) greater than 1,500/mm3, and platelets greater than 50,000/mm3
* Serum bilirubin less than 2 times the upper limit of normal range (ULN)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)
* Serum creatinine less than 2.0 times the ULN
* ECOG performance status 0, 1, 2
* Age, 20 years or older

Exclusion Criteria:

* Other malignancy, with the exception of curatively treated non-melanoma skin cancer or cervical carcinoma in situ prior to commencement of the study
* CR was confirmed more than 6 weeks prior to commencement of the study
* Concurrent treatment which may interfere with evaluation
* Pregnancy or breast feeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2008-12; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
2-year RFS | 6 years

SECONDARY OUTCOMES:
Overall survival | 8 year

CONTACTS AND LOCATIONS:
Overall Officials: Y. S. Lu, MD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan